CLINICAL TRIAL: NCT00196677
Title: Treatment of Glaucomatous Neuropathy With Food Additives
Brief Title: Study of Glaucoma Treatment With Food Additives
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial was terminated due to investigator's decision
Sponsor: Future Products Management (Other)
Responsible Party: Dr. Meir Gorban, Future Products Management
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: g88
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Glaucomatous Neuropathy
MeSH Terms: interventions — Vitamins; Minerals

INTERVENTIONS:
Drug: Vitamins, minerals and medical herbs

SUMMARY:
The purpose of this study is to determine if certain food additives are effective in the treatment of glaucoma, improving and reversing the progress of the disease.

DETAILED DESCRIPTION:
Glaucomatous neuropathy is a condition that worsens with time causing atrophy of the optic nerve and narrowing of the visual field which may culminate in blindness. The treatment tested in the trial employs certain food additives intended to reverse this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Stable open angle glaucoma - with equilibrated eye internal pressure
* Above the age of 50 years and have severe damage that does not progress to the vision field in the upper and lower half. Scoring of the vision field will be made according to the Agis study instructions.

Exclusion Criteria:

* Eye diseases excluding past cataract operation
* Allergy to one of the components in the preparation
* Deterioration in the vision field in the last year
* Kidney diseases, gastrointestinal (G.I.) tract, liver diseases, coagulation problems and thyroid diseases
* Persons who take steroids
* Diabetics or unbalanced hyperglycemia
* Autoimmune diseases
* Hypertension (not responding to treatment)
* Psychiatric treatment with drugs, psychiatric pathologies
* Pregnancy
* Ability to take more than 3 pills per day regularly
* Smoking

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Improvement in vision field (Protocol24) in a Humphrey's instrument. Scoring according to the Agis study

CONTACTS AND LOCATIONS:
Overall Officials: Meir Gorban, MD, Study Director — Future Products Management; Hani Levkovitch-Verbin, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel